CLINICAL TRIAL: NCT00166192
Title: Treatment of Melasma With Jessner's Solution vs. Trichloroacetic Acid: A Comparison of Clinical Efficacy
Brief Title: Treatment of Melasma With Jessner's Solution vs. Trichloroacetic Acid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Zakiya Rice, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024850
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Melasma
Keywords: Melasma; Jessner's solution; Trichloroacetic acid (TCA)
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemical Peel (Active Comparator): Split face treatment paradigm
  Interventions: Procedure: Jessner's solution chemical peel; Procedure: Trichloroacetic acid chemical peel

INTERVENTIONS:
Procedure: Jessner's solution chemical peel
Procedure: Trichloroacetic acid chemical peel

SUMMARY:
Melasma is an acquired discoloration of the skin characterized by brown patches. Chemical peels using agents such as Jessner's solution and trichloroacetic acid (TCA) are commonly used to treat melasma. A chemical peel involves applying the peeling agent to the skin for a short period. The skin will peel similar to a sunburn, and moisturizers are applied to the skin. Although both agents are well-accepted, there have been no good comparisons of the two agents. The purpose of this study is determine if there is a difference in the effectiveness of these two agents.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old
* Clinical diagnosis of melasma
* Mental capacity to give informed consent

Exclusion Criteria:

* Pregnancy
* H/o allergy to Jessner's solution, tricholoracetetic acid, tretinoin, or hydroquinone
* Active dermatitis
* Presence of cutaneous infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy by clinician's evaluation | 3 months
  Hyperpigmenation Global Score

SECONDARY OUTCOMES:
Efficacy by subject's evaluation | 3 months
  Hyperpigmentation Global Score

CONTACTS AND LOCATIONS:
Overall Officials: Carl Washington, MD, Principal Investigator — Emory University Department of Dermatology
Locations (1):
- Emory University Dermatology Clinic, Atlanta, Georgia, United States